CLINICAL TRIAL: NCT05124418
Title: A New Non-invasive Method to Assess and Measure Palatal Masticatory Mucosa Using Dynamic Navigation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202103099DIND
Record Dates: First submitted 2021-10-31; First posted 2021-11-18 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Palatal Masticatory Mucosa Thickness
Keywords: cone beam computed tomography,dynamic navigation,Palatal maticatory mucosa thickness,non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palatal masticatory mucosa thickness measurement (Other)
  Interventions: Diagnostic Test: palatal masticatory mucosa thickness measurement

INTERVENTIONS:
Diagnostic Test: palatal masticatory mucosa thickness measurement — Measure the thickness of palatal masticatory mucosa by a dynamic navigation system (Navident®, ClaroNav Inc., Toronto, Canada) and periodontal probe piercing.

SUMMARY:
Periodontal plastic surgery is widely used to improve the esthetic and functional demands of patients. The palatal masticatory mucosa is the main donor area. A lot of methods to evaluate the thickness of palatal soft tissue were used. However, the methods published before were invasive or non-reproducible. Therefore, the aim of this study was to investigate the accuracy of the novel invasive method to evaluate the thickness of palatal masticatory mucosa thickness.

Twelve periodontally healthy patients who will have CBCT on maxilla for implant surgery will be recruited in this study. Each patient will be measured at 15 points of palatal masticatory mucosa over canine to the second molar area, it will be done by a dynamic navigation system (test group) and periodontal probe piercing (control group). The data will be analyzed to evaluate the accuracy of dynamic navigation in the measurement of palatal masticatory mucosa thickness.

ELIGIBILITY:
Inclusion criteria:

1. Above 20 years old
2. The patient need dental implant surgery in maxilla
3. The patient have at least complete canine to second molar at one side
4. Periodontaliy healthy patients
5. The patient could sign for the consent form.

Exclusion criteria:

1. patients can not receive dental implant surgery
2. fuzzy palatal alveolar bone line
3. all maxillary posterior teeth with metal crowns
4. all posterior teeth are missing at one side over maxilla
5. all maxillary posterior teeth with hyper-mobility
6. Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
measure thickness of palatal masticatory mucosa using dynamic navigation system (in mm) and periodontal probe (in mm) | immediately after examination

SECONDARY OUTCOMES:
Information of palatal masticatory mucosa thickness in Taiwanese people | immediately after examination

CONTACTS AND LOCATIONS:
Overall Officials: CHEN-YING WANG, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan